CLINICAL TRIAL: NCT05770258
Title: A Novel Electrolyzed Water Spray Reduces the Gingival Discomfort as Well as Gingival Redness, Swelling and Bleeding of Patients With Mild Periodontitis: A Clinical Study
Brief Title: The Novel Electrolyzed Water Spray Treatment Mild Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dove Medical Press Ltd (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jia19681222
Record Dates: First submitted 2023-02-27; First posted 2023-03-15 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-02

CONDITIONS: Periodontitis
Keywords: Electrolyzed water device; Hydroxyl radical; Tap water; Spray; Periodontitis; gingival redness; gingival swelling; gingival bleeding
MeSH Terms: conditions — Periodontitis; Gingival Hemorrhage

STUDY DESIGN:
Masking Description: An open label, single arm and before and after treatment comparison study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The mild periodontitis and one treatment (Experimental): Participants with mild periodontitis accompanied by gingival discomfort will receive one treatment with the device and complete the questionnaire.
  Interventions: Device: The novel electrolyzed water spray

INTERVENTIONS:
Device: The novel electrolyzed water spray — Study staff will use the novel electrolyzed water spray device and spray for approximately 5 minutes on the participant's diseased area until half a bottle (200ml) of water is used. The patients use electrolyzed water to treat the diseased area, two times a day, for 10 days. The trial consists of 10 study visits (day 1-day 10). The relief of mild periodontitis evaluation and adverse event assessments will be performed at each visit. Safety analysis will be assessed based on the reports of adverse events during the study.

SUMMARY:
The purpose of this study is to test whether spraying the tooth of patients by use of the novel electrolyzed water spray will produce improvement in the condition of mild periodontitis.

DETAILED DESCRIPTION:
In this study, water inculding tap water,pure water and salt water, and an apparatus for producing electrolyzed water (https://www.deposon.com.cn; https://www.deposon.com）were used to generate an electrolyzed water mist spray or spray. This instantly generated electrolyzed water mist spray or spray has oxidation-reduction potential (ORP) ≥1200mv,and contains non-specific total oxidation capacity which equals to 0.28±0.10ppm,0.06±0.04ppm and 3.92±0.39ppm of desolved ozone. This instantly generated electrolyzed water mist spray or spray does not release detectable ≥0.1mg/m3 of gaseous ozone. This instantly generated electrolyzed water mist spray or spray has pH 8.4±0.4 and releases negative air ion.The apparatus for producing electrolyzed water has a positive electrode which is covered by a conductive diamond material (Patent# CN215308550U). This is an open-label, single-arm, and before and after treatment comparison study. This study uses this novel electrolyzed water device and the water spray to treat mild periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* mild periodontitis accompanied by gingival discomfort.
* Patient > 18 years old.
* Systemically healthy individuals

Exclusion Criteria:

* severe periodontitis.
* 80 years or older.
* Patients who take Anticoagulants or Antiplatelet Agents
* Pregnant or breastfeeding women

Ages: 36 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-29 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
A discomfort or itching scale made by modifying the Numeric Pain Rating Scale (NPRS) | 10 days
  This Score is based on descriptions of the itching that patients rate 0-10 to assess the condition of their gingival with itching. A higher score means a worse outcome. 0 means "no itching " and 10 means "the most itching".

SECONDARY OUTCOMES:
A gingival signs scale made by modifying the Numeric Pain Rating Scale (NPRS). | 10 days
  A gingival signs scale evaluates the signs of gingival redness, swelling and bleeding in patients with mild periodontitis. This Score is based on descriptions of signs of gingival redness, swelling and bleeding with patients rated 0-10 to assess the condition of mild periodontitis. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Huinuode Biotechnology Co., Ltd., Qingdao, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: until publication of this clinical study and international patent granted